CLINICAL TRIAL: NCT03118583
Title: An Open-label, Pilot Trial to Assess the Effects of a Dietary Supplement on Fasting Lipoprotein Lipids and a Marker of Inflammation in Men and Women With Above-desirable Levels of Low-density Lipoprotein Cholesterol
Brief Title: Effects of a Dietary Supplement on Lipoprotein Lipids and Inflammatory Markers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Midwest Center for Metabolic and Cardiovascular Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MB-1608
Record Dates: First submitted 2017-04-08; First posted 2017-04-18 (Actual); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dietary supplement with carrageenan (Experimental): 300 mg/day of dietary supplement containing carrageenan
  Interventions: Dietary Supplement: 300 mg/day of dietary supplement containing carrageenan

INTERVENTIONS:
Dietary Supplement: 300 mg/day of dietary supplement containing carrageenan — 300 mg/day of dietary supplement containing carrageenan.

SUMMARY:
The goal of this study is to assess the effects of a dietary supplement on fasting lipoprotein lipids and a marker of inflammation in men and women with levels of low-density lipoprotein cholesterol above desirable levels.

DETAILED DESCRIPTION:
Carrageenan is a naturally occurring plant polysaccharide extracted from edible seaweeds that is widely used in food and beverage products, with a history of use dating back hundreds of years. It is an FDA-approved food additive in the U.S. and has regulatory approval for use as a food ingredient in Europe, Asia, and Latin America.

An earlier clinical trial conducted by the Russian Academy of Sciences demonstrated that consumption of 250 mg/day of carrageenan in capsules, for 28 days, lowered low-density lipoprotein cholesterol (LDL-C) by 34%. In that study, carrageenan consumption also resulted in statistically significant decreases in important biomarkers of chronic inflammation: leukocytes by 16%, fibrinogen by 9%, and C-reactive protein (CRP) by 13%. Another clinical trial conducted by the University of the Philippines showed that carrageenan added to foods led to statistically significant decreases in total cholesterol (total-C) and triglycerides (TG), elevated levels of which are also linked to cardiovascular disease. That study showed that carrageenan consumption led to a 33% reduction in total-C and a 32% reduction in TG.

This is a pilot, open-label, 4 week trial with two screening visits, one baseline visit and two test visits. Subjects will consume 300 mg/day of a proprietary dietary capsule containing carrageenan, with a meal at a consistent time each day, starting at the baseline visit. Fasting blood samples will be collected for lipid profile (total-C, LDL-C, high-density lipoprotein cholesterol [HDL-C], and TG), and high-sensitivity CRP (hs-CRP) measurements at the second screening visit, baseline and the two test visits. Additionally, blood will be drawn for a comprehensive metabolic panel and complete blood count at the second screening and the last test visit only. Assessments of vital signs, body weight, evaluation of inclusion and exclusion criteria, concomitant medication/supplement use, and adverse events will be performed throughout the study. Written study instructions will be provided to the subjects including instructions about fasting, maintenance of adequate hydration, and refraining from vigorous physical activity, alcohol consumption, and tobacco products prior to and during the subsequent visit. At the end of the 4 week test period, subjects will return study product and compliance will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index 18.5-34.9 kg/m2
2. Judged to be in good health on basis of medical history and screening laboratory tests
3. Fasting LDL-C ≥115 mg/dL and <190 mg/dL

Exclusion Criteria:

1. Abnormal laboratory test results of clinical significance (e.g., TG ≥400 mg/dL, blood glucose ≥126 mg/dL, fasting creatinine ≥1.5 mg/dL, alanine aminotransferase or aspartate aminotransferase ≥1.5X the upper limit of normal)
2. Atherosclerotic cardiovascular disease or other evidence of atherosclerotic cardiovascular disease (myocardial infarction or other acute coronary syndrome, coronary or other revascularization procedure, transient ischemic attack, ischemic stroke, atherosclerotic peripheral arterial disease or other documented atherosclerotic diseases)
3. Recent major trauma or surgical event
4. History or presence of clinically important pulmonary, endocrine, hepatic, renal, hematologic, immunologic, dermatologic, neurologic, psychiatric, or biliary disorders
5. History or current gastrointestinal disorder with the potential to disrupt normal digestion and absorption
6. Known allergy, sensitivity, or intolerance to any ingredients in the study product
7. Uncontrolled hypertension
8. Recent history of cancer (except non-melanoma skin cancer)
9. Recent weight change ≥4.5 kg
10. History of diagnosed eating disorder
11. Extreme dietary habits
12. Current or recent history of, or strong potential for, drug or alcohol abuse
13. Recent use of medications intended to alter the lipid profile, (e.g., statins, bile acid sequestrants, cholesterol absorption inhibitor, fibrates, niacin [drug form] or omega-3 fatty acid drugs), weight-loss drugs or programs, systemic corticosteroids, anticoagulants, or unstable use of any antihypertensive medication
14. Recent use of foods or dietary supplements with potential to influence lipid metabolism (e.g., omega-3 fatty acid supplements or fortified foods, sterol/stanol products, red rice yeast supplements, garlic supplements, soy isoflavone supplements, niacin or its analogues at doses >400 mg/d) and viscous dietary fiber supplements (e.g., psyllium, beta-glucan, methylceullylose and/or carrageenan)
15. Recent use of antibiotics
16. Pregnant, planning to be pregnant during the study period or lactating females or women of childbearing potential unwilling to commit to use of a medically approved form of contraception

Ages: 25 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
LDL-C | Up to 28 days
  Percent change in LDL-C from baseline (average of values at days -7 and 0) to end of treatment (average of values at days 21 and 28)

SECONDARY OUTCOMES:
Total-C | Up to 28 days
  Percent change in total-C from baseline (average of values at days -7 and 0) to end of treatment (average of values at days 21 and 28)
HDL-C | Upto 28 days
  Percent change in HDL-C from baseline (average of values at days -7 and 0) to end of treatment (average of values at days 21 and 28)
Total-C/HDL-C | Up to 28 days
  Percent change in the ratio of total-C/HDL-C from baseline (average of values at days -7 and 0) to end of treatment (average of values at days 21 and 28)
Non-high-density lipoprotein cholesterol (non-HDL-C) | Upto 28 days
  Percent change in non-HDL-C (calculated as total-C minus HDL-C) from baseline (average of values at days -7 and 0) to end of treatment (average of values at days 21 and 28)
Triglycerides (TG) | Up to 28 days
  Percent change in TG from baseline (average of values at days -7 and 0) to end of treatment (average of values at days 21 and 28)
hs-CRP | Up to 28 days
  Change in hs-CRP from baseline (average of values at days -7 and 0) to end of treatment (average of values at days 21 and 28)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin C Maki, PhD, Study Director — MB Clinical Research and Consulting LLC
Locations (1):
- MB Clinical Research, Boca Raton, Florida, United States

IPD SHARING:
Plan to Share IPD: No